CLINICAL TRIAL: NCT04811859
Title: The Effect of Inspiratory Muscle Training on Respiratory Muscle Strength, Respiratory Functions and Functional Capacity in Post COVID-19 Patients
Brief Title: The Effect of Inspiratory Muscle Training in Post COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISUCPR
Record Dates: First submitted 2021-02-25; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Infective Pneumonia
Keywords: Inspiratory Muscle Training; Post-COVID 19; Respiratory Muscle Strength; Respiratory Function; Functional Capacity
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): In the study group, Inspiratory Muscle Training will be applied with Threshold IMT device (Respironics, USA) at 40% of the maximum inspiratory pressure value for eight weeks, every day of the week, twice a day for 15 minutes. The patients will come for a control once a week, the maximum inspiratory pressure will be measured again and the new training intensity will be determined at 40% of the new maximum inspiratory pressure.
  Interventions: Other: Inspiratory Muscle Training
- Control group (Sham Comparator): In the control group, Inspiratory Muscle Training will be applied with Threshold IMT device (Respironics, USA) at 10% of the maximum inspiratory pressure value for eight weeks, every day of the week, twice a day for 15 minutes. The exercise workload will not be increased and will remain the same. It will run at 10% of maximum inspiratory pressure for eight weeks.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory Muscle Training is a form of resistance (weight) training which strengthens the muscles that you use to breathe. When these muscles are strengthened regularly for a period of a few weeks they adapt, becoming stronger and being able to work for longer.

SUMMARY:
The COVID-19 infection, which is considered as a pandemic by the World Health Organization, affects the whole world. COVID-19 is an infectious respiratory disease caused by SARS-CoV-2. It is stated in early studies that after COVID-19 infection, there are adverse effects on both the peripheral and respiratory muscles along with the pulmonary system involvement. The purpose of our study; To examine the effect of Inspiratory Muscle Training (IMT) on respiratory muscle strength, respiratory functions and functional capacity in PostCOVID-19 patients. Patients who have been hospitalized and discharged with the diagnosis of COVID-19 in Istinye University hospitals, at least 6 weeks have passed since the infection, the PCR test has turned negative will be taken. The evaluation and treatment of the patients will be carried out in the Education and Research Units of Istinye University Physiotherapy and Rehabilitation Department. Patients included in the study will be randomly divided into two groups, study and control groups. Demographic evaluation form, Post Covid Functional Status Scale, Charlson Comorbidity Index, Modified Medical Research Council (MMRC) Dyspnea scale, Corbin posture analysis, Respiratory function test, Respiratory muscle strength measurement, Respiratory Muscle Endurance measurement, 6-minute walking test (6 MWT) ), Peripheral Muscle Strength, Grip Strength, Hospital Anxiety and Depression Scale (HADS), Breathlessness Perception Questionnaire (BBQ) and Nottingham Health Profile Questionnaire will be used. In the study group, IMT will be applied at 40% of the maximum inspiratory pressure (MIP) for eight weeks, every day of the week, twice a day for 15 minutes. The patients will come for a control once a week, the MIP values will be measured again and the new training intensity will be determined at 40% of the new MIP value. The control group will be given a constant training of 15 minutes at 10% of the MIP, twice a day, every day of the week for eight weeks. Evaluations of the study and control groups will be made at the beginning and after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-70
* Being clinically stable,
* Having COVID-19 infection and at least 6 weeks after infection
* Being between Grade 2-4 according to Post-COVID Functional Status Scale
* Regular participation in treatment
* To read, write and understand Turkish
* Volunteering to participate in research

Exclusion Criteria:

* Presence of mental and cognitive impairments
* Having an orthopedic, neurological disease that prevents exercise
* Uncontrolled hypertension, having a cardiovascular disease
* Pregnancy and breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
PostCovid Functional Status Scale | eight weeks
  PostCovid Functional Status Scale: It will be used to assess the functional status of patients after COVID-19 infection. It divides the functional status of the patients into stages between 0 and 4.
Pulmonary Function Test | eight weeks
  Pulmonary Function Test will be performed using a portable spirometry according to the guidelines of the American Thoracic Society. Forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC), and peak expiratory flow (PEF) will be expressed as the percentages of the predicted values.
Inspiratory muscle strength | eight weeks
  Inspiratory muscle strength are the static inspiratory pressure measured at the mouth. It is called maximal inspiratory pressure (MIP) and it will be assessed using an electronic pressure transducer. The MIP will be measured at residual volume.
Functional capacity | eight weeks
  Six-minute walk test (6MWT) will be applied in a 30-m unobstructed corridor. Patients and controls will be instructed to walk their own pace but to cover as much meter as possible within 6 min.The distance will be recorded.
Expiratory muscle strength | eight weeks
  Expiratory muscle strength are the static expiratory pressure measured at the mouth. It is called maximal expiratory pressure (MEP) and it will be assessed using an electronic pressure transducer. The MEP will be measured from total lung capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No